CLINICAL TRIAL: NCT02522195
Title: Meal Distribution Across the Day in Female Nurses Working Shifts and Their Relationship With Nutritional Status
Brief Title: Meal Distribution Across the Day in Female Nurses Working Shifts
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Martina Pafume Coelho, MsC, Federal University of Uberlandia
Other Study IDs: FUUberlandia
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder; Imbalance of Constituents of Food Intake
Keywords: shift work; nutritional status; nursing professionals; meal distribution; food intake

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study assessed the meal distribution across the day (energy and macronutrient intake) and its relationship to the nutritional status of nursing professionals.

DETAILED DESCRIPTION:
221 female nursing professionals from Brazilian University hospital were classified in three shifts: day shift (n=112), night shift (n=55), and day-night shift (n=54).

Food intake assessment (3-day 24-hour recall); Anthropometric variables (weight, height, waist circumference and hip circumference); Sleep time on working days and day off.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were regularly employed by the hospital, with 36-hours per week scheduke, not counting additional shifts and overtime work.

Exclusion Criteria:

* Volunteers who did not supply the necessary information for the development of the research and who were pregnant or lactating.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Woman who were part of Nursing Staff of University Hospital, and agreed to participate in the study. Each volunteer provided a full, written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
meal distribution | 1 year
  3-Day 24-Hour Recall Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Cibele Crispim, PhD, Principal Investigator — Federal University of Uberlandia